CLINICAL TRIAL: NCT04289454
Title: Ketone Esters for Optimization of Operator Performance in Hypoxia Technical Volume (Sub-project: Sensory Analysis and Taste Modulation of the Ketone Ester)
Brief Title: Sensory Analysis and Taste Modulation of Ketone Esters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Monell Chemical Senses Center (Other)
Collaborators: HVMN (funding; holder of primary Department of Defense STTR contract) (Unknown)
Responsible Party: Principal Investigator, Paul Wise, Associate Member (equivalent to Associate Professor), Monell Chemical Senses Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SUB055AO1PWise; H92405-19-C-0016 (Other Grant/Funding Number: SOCOM)
Record Dates: First submitted 2020-02-18; First posted 2020-02-28 (Actual); Last update posted 2022-03-21 (Actual); Status verified 2022-03

CONDITIONS: Flavor Perception in Normal, Healthy Adults
MeSH Terms: interventions — Flavoring Agents

STUDY DESIGN:
Intervention Model Description: Within-subjects design (the same group of subjects will taste model KE drinks with vs. without added flavors), with order counter-balanced.
Masking Description: Samples presented will not be identified (there will be no codes or visual cues regarding whether a model drink does or does not contain a flavor modifier). However, true blinding is impossible since flavor will differ between samples.
  Investigators will not be blind to sample contents. However, responses will be collected and recorded using an automated computer program, which offers some protection against possible experimenter bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Effect of flavor modifiers (Other): Intervention in the study: Subjects will taste model KE drinks with (control condition) and without (experimental condition) added flavors. Design is within-subjects (subjects will taste both the experimental and control drinks), with order counter-balanced across subjects.
  Interventions: Other: Flavor additive

INTERVENTIONS:
Other: Flavor additive — Various flavor additives will be tested (vs. no added flavor) to determine which show promise for making KE drinks taste less unpleasant

SUMMARY:
Ketone ester (KE) drinks are sold commercially in the USA and elsewhere (the FDA has accepted a GRAS (generally regarded as safe) notification on the KEs we propose to study). KE drinks can have beneficial effects on metabolism. Unfortunately, KE drinks have a strongly unpleasant flavor which can trigger rejection. The current study will generate data to help inform KE drink formulations with improved flavor. First stage, trained subjects will rate the intensity of various sensation qualities (e.g., bitter, sour, metallic, and astringent) from KE drinks to help understand the nature of the unpleasant flavor and the particular sensory systems involved (e.g., taste vs. smell). Then, subjects will taste KE drinks with and without various flavor modifiers. Subjects will be healthy adults (aged 21-45) without known food allergies.

ELIGIBILITY:
Inclusion Criteria:

1. Good general health (self report)
2. Men and women
3. Age from 21 to 45

Exclusion Criteria:

1. Current (or within the last four weeks) acute illness, such as cold or flu
2. Currently active allergies
3. Regular use of medication (over the counter or prescription), except for birth control.
4. Any history of food allergy or sensitivity (particularly to KE drinks or MSG). Any history of sensitivity to 6-Propylthiouracil (bitter compound frequently used to assess individual differences in sensitivity to bitterness).
5. Pregnant, nursing, or trying to become pregnant during the study (pregnancy can affect flavor perception)
6. Chronic illness (any ongoing condition that is serious or required medical monitoring), including kidney problems, liver problems, cardiovascular problems (e.g., heart disease or high blood pressure), diabetes, HIV infection, or other ongoing illness). Diabetes or other metabolic issues could be important for safety as well as quality of data.
7. History of taste problems (absent or abnormal sense of taste)
8. Weigh less than 100 pounds (45.4 kilograms). This is to help ensure that the amount of KE drink consumed remains below the single serving in the GRAS (generally regarded as safe) notice which the FDA has accepted.

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2020-08-30 (Actual); Primary Completion 2021-06-04 (Actual); Study Completion 2021-06-04 (Actual)

PRIMARY OUTCOMES:
Rated intensity profile | Through study completion (up to a year for a given participant, depending on how many drink samples the participant agrees to evaluate). Participants will rate the intensity of about 12 model drink samples during each study visit.
  Rated intensity of taste qualities (e.g., sour, bitter) and mouth-feel (astringent) of model drinks, measured using the general Labeled Magnitude Scale (gLMS). In this implementation of the gLMS, scores will range from 0 (or "no sensation") up to 100 ("strongest imaginable sensation"), with higher scores indicating stronger perceived intensity for the sensation in question.

SECONDARY OUTCOMES:
Hedonic response | Through study completion (up to a year for a given participant, depending on how many drink samples the participant agrees to evaluate). Participants will rate the pleasantness of about 12 model drink samples during each study visit.
  Ratings of how likely the flavor of each sample tasted would be to discourage use of a product with that flavor, assuming the rater otherwise wanted associated nutritional or performance benefits
Rated upper GI symptoms | Through study completion (up to a year for a given participant, depending on how many drink samples the participant agrees to evaluate). Participants will rate upper GI symptoms after tasting about 12 model drink samples during each study visit.
  Rated intensity of nausea, bloating, and heartburn, using a nine-point category scale (some bitter liquids can trigger mild to moderate feelings of nausea). Scores for each symptom range from 0 ("none") to 8 ("Unbearable"), with "mild" (2), "moderate" (4), and "severe" (6) as labeled intermediate categories.

CONTACTS AND LOCATIONS:
Overall Officials: Paul M Wise, PhD, Principal Investigator — Monell Chemical Senses Center
Locations (1):
- Monell Chemical Senses Center, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided
If individual subject data are shared, the data will be de-identified first (no identifying information will be shared with other researchers).

DOCUMENTS (1):
  • Informed Consent Form (2022-01-19): https://cdn.clinicaltrials.gov/large-docs/54/NCT04289454/ICF_001.pdf